CLINICAL TRIAL: NCT06934980
Title: A PHASE 0, EVALUATION OF MICRONEEDLE-BASED COLLECTION OF DERMAL INTERSTITIAL SKIN FLUID IN HEALTHY PARTICIPANTS AND ATOPIC DERMATITIS PATIENTS
Brief Title: A Study to Evaluate Microneedle-based Collection of Dermal Interstitial Skin Fluid in Healthy Participants and Atopic Dermatitis Participants
Status: Completed | Type: Observational
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INCB000000-002
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis; Healthy Volunteers
Keywords: Microneedle Device
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collecting biospecimens (dermal interstitial skin fluid (dISF), blood, skin tape strip, and biopsy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Healthy Volunteers: Microneedle device samples will be collected as defined in the protocol as a non-invasive method.
  Interventions: Device: Microneedle Device
- Participants with Atopic Dermatitis (AD): Microneedle device samples will be collected as defined in the protocol as a non-invasive method.
  Interventions: Device: Microneedle Device

INTERVENTIONS:
Device: Microneedle Device — Microneedle device will be used for collecting dermal interstitial skin fluid samples as defined by the protocol.

SUMMARY:
The purpose of this study is to evaluate microneedle-based collection of dermal interstitial skin fluid (dISF) in healthy participants and atopic dermatitis (AD) participants

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Male or female participant aged 18 to 65 years (inclusive) at the time of consent.
* Female participant of childbearing potential has a negative urine pregnancy test at screening and Day 1.
* Participant is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
* Participants must be willing and able to comply with all study procedures and must be available for the duration of the study.

Healthy Participants:

* Participant is in good general health, according to the investigator's judgment based on medical and surgical history and skin examination.
* Participant has no known prior history of autoimmune inflammatory skin conditions.

Participants with AD:

* Participant has clinically confirmed diagnosis of active AD, according to Hanifin and Rajka criteria.
* Participant has at least 2 years history of AD (information obtained from medical chart or participant's physician, or directly from the participant) and had no significant flares in AD for at least 4 weeks before screening according to investigators judgement.
* Participant has mild to severe AD at screening and Day 1, as defined by an IGA ≥ 2.
* Participant has AD covering ≥ 3% of the BSA (excluding palms, soles, scalp, genitals, and folds) at screening and Day 1.
* Participant has ≥ 2 target lesions with a TLSS score ≥ 6 at screening and Day 1 (Lesion Sites #1 and #2) with a lesional surface allowing the collection of all required biospecimens. The difference in TLSS between the 2 target lesions must not be > 1.

Note 1: A participant who does not have a Lesion Site #2 with a lesional surface that could accommodate all biospecimens collection may be enrolled in the study if he/she has individual AD lesions (collectively referred to as Lesion Site #2) amenable to sample collection that have (1) an overall surface to accommodate all biospecimens collection, (2) identical TLSS scores, and are (3) from the same anatomical region.

Note 2: Every effort should be made to collect all required biospecimens at Lesion Site #2. However, if lesional size does not allow, the tape strip sample may not be collected. A minimum of 8 patients with AD should undergo tape strip sample collection at Lesion Site #2.

Exclusion Criteria:

All Participants:

* Participant is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Participant is known to have immune deficiency or is immunocompromized.
* Participant has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Participants with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
* Participant had a major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
* Participant has a known history of clinically significant drug or alcohol abuse in the last year prior to Day 1.
* Participant has received an investigational product or device within 4 weeks or 5 half-lives (whichever is longer) prior to Day 1.
* Participant has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.
* Participant has a presence of any tattoos, scratches, open sores, excessive hair, or skin damage that, in the opinion of the investigator, may interfere with study evaluations.
* Participant is unlikely, in the opinion of the investigator, to be compliant with study procedures and requirements.
* Participant has a close affiliation (eg, a close relative) with the investigator, including any study staff of the sites or persons working at the contract research organization, or participant is an employee of the sponsor.
* Participant has a known history of chronic infectious disease (eg, hepatitis B, hepatitis C, or human immunodeficiency virus [HIV]).
* Participant has had excessive sun exposure, is planning a trip to a sunny climate, or has used tanning booths within 4 weeks prior to Day 1. Use of sunscreen products and protective apparel are recommended when sun exposure cannot be avoided.
* Participant is institutionalized because of legal or regulatory order.
* Participant has used any topical product in the sampling area prior to the visit on Day 1.
* Participant has received a live or live-attenuated vaccine within 4 weeks prior to Day 1.

Healthy Participants:

* Participant has used topical medication (prescription or over-the-counter [OTC]) in the sampling area within 2 weeks prior to Day 1.
* Participant has used prescription immunosuppressive or immunomodulatory drugs within 4 weeks prior to Day 1.

Participants with AD:

* Participant has clinically infected AD.
* Participant has any clinically significant medical condition abnormality (based on medical and surgical history and skin examination) that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of study results.
* Participant has used doxepin within 1 week prior to Day 1.
* Participant has used hydroxyzine or diphenhydramine within 1 week prior to Day 1.
* Participant has used topical products containing urea within 1 week prior to Day 1.
* Participant has used systemic antibiotics within 2 weeks or topical antibiotics within 1 week prior to Day 1.
* Participant has used any topical medicated treatment that could affect AD within 1 week prior to Day 1, including, but not limited to, topical corticosteroids, crisaborole, calcineurin inhibitors, ruxolitinib, tars, antimicrobials, medical devices, and bleach baths.
* Participant has used systemic treatments (other than biologics) that could affect AD less than 4 weeks prior to Day 1, including, but not limited to, retinoids, calcineurin inhibitors, methotrexate, cyclosporine, azathioprine, oral/injectable corticosteroids, baricitinib, upadacitinib, and abrocitinib.

Note: Intranasal corticosteroids and inhaled corticosteroids are allowed. Eye and ear drops containing corticosteroids are also allowed.

* Participant has received any ultraviolet (UV)-B phototherapy (including tanning beds) or excimer laser within 4 weeks prior to Day 1.
* Participant has had psoralen-UV-A (PUVA) treatment within 4 weeks prior to Day 1.
* Participant has received any marketed (eg, dupilumab, tralokinumab, lebrikizumab) or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
* Participant has received an intravenous immunoglobulin (IVIg) therapy within 12 weeks prior to Day 1.
* Participant has a history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
* Participant has a history of hypertrophic scarring or keloid formation in scars or suture sites.
* Participant has taken anticoagulant medication, such as heparin, low molecular weight (LMW)-heparin, warfarin, antiplatelets (except low-dose aspirin ≤ 81 mg which will be allowed), within 2 weeks prior to Day 1, or has a contraindication to skin biopsies. Nonsteroidal anti-inflammatory drugs (NSAIDs) will not be considered antiplatelets and will be allowed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 5 healthy participants and approximately 10 to 15 participants with mild to severe AD will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Volume of dISF collected from normal skin in healthy participants and lesional skin from AD patients | Day 1

SECONDARY OUTCOMES:
Incidence and severity of procedural complications | Up to 14 days
  Defined using the Investigator Global Assessment Scale.
Willingness for repeat sample collection | Day 1
  Defined using a 5- point likert scale questionnaire.
Tolerability of dISF collection and other sampling techniques | Day 1
  Defined using the Local Skin Tolerability Scale.
Tolerability of a single and two consecutive dISF sample collection in a single day | Day 1
  Defined using the Local Skin Tolerability Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate Microneedle-based Collection of Dermal Interstitial Skin Fluid in Healthy Participants and Atopic Dermatitis Participants — https://incyteclinicaltrials.com/studies/incb000000-002